CLINICAL TRIAL: NCT06584383
Title: Early Focus II: A Prospective, Randomized, Controlled Trial to Test Safety and Effectiveness of Unilateral Exablate MR-guided Focused Ultrasound (MRgFUS) Subthalamotomy in Patients With Early-Stage Parkinson's Disease (ESPD)
Brief Title: A Prospective, Randomized, Controlled Trial to Test Safety and Effectiveness of Unilateral Exablate MR-guided Focused Ultrasound Subthalamotomy in Patients With Early-Stage Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD017
Record Dates: First submitted 2024-08-30; First posted 2024-09-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Exablate; MRgFUS; Subthalamotomy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: It is contemplated that, if the patients from the control arm require unilateral Exablate MRgFUS subthalamotomy, the treatment could be performed after Month 12 visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exablate Arm (Experimental): Subjects will receive Exablate MRgFUS subthalamotomy
  Interventions: Procedure: Exablate MRgFUS subthalamotomy
- Control Arm (Active Comparator): Subjects will receive best medical treatment. It is contemplated that, if the patients from the control arm require unilateral Exablate MRgFUS subthalamotomy, the treatment could be performed after Month 12 visit.
  Interventions: Procedure: Exablate MRgFUS subthalamotomy; Drug: Best Medical Treatment
- Reference Arm (Active Comparator): Patients fulfilling all inclusion/exclusion criteria except for the SDR requirements (and so anatomically not able to undergo MRgFUS subthalamotomy) will be offered the option to receive best medical treatment and will be formally followed as a reference comparator for up to 3 years.
  Interventions: Drug: Best Medical Treatment

INTERVENTIONS:
Procedure: Exablate MRgFUS subthalamotomy — Exablate MRgFUS subthalamotomy for Parkinson's Disease
  Arms: Control Arm; Exablate Arm
Drug: Best Medical Treatment — Subjects will be managed according to conventional therapeutic guidelines (i.e., best medical treatment) for Parkinson's Disease
  Arms: Control Arm; Reference Arm

SUMMARY:
This prospective, randomized, multicenter study aims to evaluate in Early-Stage Parkinson's Disease (ESPD) patients the safety and effectiveness of treatment with Exablate MRgFUS subthalamotomy vs best medical treatment.

DETAILED DESCRIPTION:
This is a prospective, randomized (ratio 2:1), multicenter study to evaluate in Early-Stage Parkinson's Disease (ESPD) patients the safety and effectiveness of treatment with Exablate MRgFUS subthalamotomy vs best medical treatment. Patients assigned to the treatment arm will receive unilateral Exablate MRgFUS subthalamotomy. Patients assigned to control group will receive best medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women; age 30 to 65 years old
* Subjects who are able and willing to give consent and able to attend all study visits. - Subjects with a diagnosis of PD according to the modified clinical criteria by the Movement Disorders Society, for less than 5 years and more than 12 months.
* Off-medication MDS-UPDRS part III of the most affected body side ≥ 10
* Motor signs predominantly present in one body side: Asymmetry index (MDS-UPDRS III of the most affected side/MDS-UPDRS III of the least effected side) ≥ 2.
* Patients should have a stable pharmacological regime for the last 4-weeks prior to baseline evaluation.
* Topographic coordinates of the subthalamic nucleus are localizable on MRI so that it can be targeted by the Exablate device.
* Skull density ratio (SDR) score of 0.40 or higher*. The SDR is a determinant factor for the suitability to MRgFUS ablation. SDR is a ratio of ultrasound energy penetration through the skull. The SDR threshold for using Exablate 4000 is established at 0.4 with patients having SDR below that value considered unsuitable candidates.
* Able to communicate sensations during the Exablate MRgFUS treatment.

Exclusion Criteria:

* MDS-UPDRS part III OFF medications > 32 in the off state and/or Hoehn and Yahr state ON medication greater than 2.
* Significative evidence (by clinical history) of having developed features indicative of PD motor onset 2 or more years prior to formal diagnosis.
* Presence of clinically relevant levodopa-induced dyskinesia and/or motor fluctuations as noted by a score > 1 on questions 4.2 or 4.4 of the MDS-UPDRS, that assess disability resulting from motor complications.
* Levodopa daily dose higher than 500mg or 750 levodopa-equivalents daily.
* Presence of any symptoms or signs suggesting other central neurodegenerative disease such as multisystem atrophy, progressive supranuclear palsy, cortico-basal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
* Any suspicion that parkinsonian symptoms are a side effect attributable to intake of neuroleptic or other medications.
* Subjects who have had deep brain stimulation or a prior stereotactic ablation for the treatment of movement disorders.
* Presence of significant cognitive impairment measured by standard of care method at the center.
* Patients with clinically relevant co-morbidity such as severe hypertension, diabetes, cardiac, metabolic, and psychiatric conditions
* Other exclusion criteria for the Exablate system.
* Subjects with significant depression as determined following a comprehensive assessment by a neuropsychologist. Significant depression is being defined quantitatively as a score of greater than 14 on the Beck Depression Inventory.
* Legal incapacity or limited legal capacity as determined by the neuropsychologist.
* Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within the preceding 12-month period:

  * Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
  * Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use).
  * Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct).
  * Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
* Subjects with unstable cardiac status including:

  * Unstable angina pectoris on medication
  * Subjects with documented myocardial infarction within six months of protocol entry
  * Significant congestive heart failure defined with ejection fraction <40.
  * Subjects with unstable ventricular arrhythmias
  * Subjects with atrial arrhythmias that are not rate controlled.
  * Severe hypertension (diastolic BP >100 on medication).
* History of or current medical condition resulting in abnormal bleeding and/or coagulopathy.
* Receiving anticoagulant (e.g., warfarin) or antiplatelet (e.g., aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g., Avastin) within one month of focused ultrasound procedure.
* Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard.
* Patient with severely impaired renal function with estimated glomerular filtration rate <30mL/min/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis.
* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Significant claustrophobia that cannot be managed with mild medication.
* Subject who weighs more than the upper weight limit of the MR table and who cannot fit into the MR scanner.
* Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
* History of intracranial hemorrhage.
* History of multiple strokes, or a stroke within past 6 months.
* Subjects with a history of seizures within the past year.
* Subjects with malignant brain tumors.
* Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment.
* Any illness that in the investigator's opinion preclude participation in this study.
* Subjects unable to communicate with the investigator and staff.
* Pregnancy or lactation.
* Patients without clinically relevant parkinsonism in the off- state as evaluated by two examining neurologists (or MDS- UPDRS III in the most affected side <10).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS Part III OFF Medication | 12 Months
  Between-group difference in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III at 12 months in the off-medication state.

SECONDARY OUTCOMES:
PD-specific spatial covariance patterns (PDRP or PD related metabolic pattern) with brain 18F-fluorodeoxyglucose- Positron emission tomography | 12 Months
  The metabolic pattern will be quantified to obtain a PDRP expression scores at baseline, 12-month and to compare disease evolution between groups.
MDS-UPDRS III OFF-med video-based evaluation | 12 Months
  Between group comparison through month 12 and within group comparison vs baseline month 12 in MDS-UPDRS III OFF-med video-based evaluation by a blinded movement disorders neurologist (only at baseline and 12 months).
MDS-UPDRS I, II, III (ON and OFF meds) and UPDRS IV | 12 Months, 24 Months, 36 Months
  Between group comparison through month 12 and within group comparison vs baseline month 12 to 36 in MDS-UPDRS I, II, III (ON and OFF meds) and UPDRS IV
MDS Unified Dyskinesia Rating Scale | 12 Months, 24 Months, 36 Months
  Between group comparison through month 12 and within group comparison vs baseline month 12 to 36 in MDS Unified Dyskinesia Rating Scale
Quality of life assessment (PDQ39) | 12 Months, 24 Months, 36 Months
  Between group comparison through month 12 and within group comparison vs baseline month 12 to 36 in Quality-of-life assessment (PDQ39)
Medication change | 12 Months, 24 Months, 36 Months
  Between group comparison through month 12 and within group comparison vs baseline month 12 to 36 in Parkinson's Disease medication change
MDS-Non motor rating scale | 12 Months, 24 Months, 36 Months
  Between group comparison through month 12 and within group comparison vs baseline month 12 to 36 in MDS-Non motor rating scale
Patient Global Impression of Change (PGIC) | 12 Months, 24 Months, 36 Months
  Between group comparison through month 12 and within group comparison vs baseline month 12 to 30 in Patient Global Impression of Change (PGIC)
Clinician Global Impression of Change (CGIC) | 12 Months, 24 Months, 36 Months
  Between group comparison through month 12 and within group comparison vs baseline month 12 to 30 in Clinician Global Impression of Change (PGIC)

OTHER OUTCOMES:
Safety: Incidence and frequency of adverse events related to the treatment. | 36 Months
  Incidence and frequency of adverse events related to the treatment. The investigator will capture any untoward events related to the treatment in the case report forms along with severity, duration, and resolution, and whether the event is considered serious. The severity of adverse events will be categorized according to the definition of adverse events from the International Organization for Standardization (ISO).
Exploratory assessment: F- Dopa PET assessment | 12 Months, 36 Months
  F- Dopa PET assessment will evaluate difference in the progression of striatal dopaminergic denervation.
Exploratory assessment: Time to Parkinson's Disease Progression | 12 Months, 24 Months, 36 Months
  PD progression will also be defined by comparing between-group Kaplan-Meier curves of subjects exceeding the worsening thresholds of specific clinical scales

CONTACTS AND LOCATIONS:
Overall Officials: José Obeso, MD, PhD, Principal Investigator — HM CINAC- Hospital Universitario HM Puerta del Sur; Raúl Martínez-Fernández, MD, PhD, Principal Investigator — HM CINAC- Hospital Universitario HM Puerta del Sur
Locations (4):
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Universitätsklinikum Schleswig-Holstein, Campus Kiel (UKSH), Kiel, Germany
- Spain (2):
  - HM CINAC- Hospital Universitario HM Puerta del Sur, Móstoles
  - Clinica Universidad de Navarra, Pamplona